CLINICAL TRIAL: NCT04832412
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Study of the Effect of BrainPhyt on Cognitive Function in Healthy Older Subjects
Brief Title: Effect of BrainPhyt, a Microalgae Based Ingredient on Cognitive Function in Healthy Older Subjects
Acronym: PHAEOSOL-THREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microphyt (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-126
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Healthy Aging; Dietary Supplement; Fucoxanthin; Cognitive Impairment; Neuroprotection; Mood; Stress; Sleep
MeSH Terms: conditions — Cognitive Dysfunction | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrainPhyt Low dose (Experimental): 2 capsules of 275mg BrainPhyt for 24 weeks
  Interventions: Dietary Supplement: BrainPhyt
- Placebo (Placebo Comparator): 2 capsules of 275mg Maltodextrin
  Interventions: Dietary Supplement: 100 % Maltodextrin

INTERVENTIONS:
Dietary Supplement: BrainPhyt — BrainPhyt low dose supplementation during 6 months
  Arms: BrainPhyt Low dose
Dietary Supplement: 100 % Maltodextrin — 100 % Maltodextrin
  Arms: Placebo

SUMMARY:
In developed countries, the acceleration of the general population ageing has been widely described for decades, involving changes in public health policies. Among the health issues arising from this demographic change, the maintenance of cognitive function will be a major challenge in the next years, both in societal and economic terms. In this regard, some pharmacological and behavioural (e.g. physical activity, social involvement, intellectually demanding activities) preventive approaches have been evaluated to improve cognitive function with ageing. Among them, dietary interventions showed a potential interest to prevent cognitive decline during ageing. In this sense, there is a growing interest to find ecological solutions and to meet major societal challenge the use of microalgae as molecule of interest sources is a recent promising approach. Marine environments harbour a huge biological diversity of microalgae that represents a large source of almost untapped bioactive compounds. This biodiversity comprises 200,000 to 2 million species with about 35,000 which are described and 15,000 maintained in culture collections. Microalgae are able to produce bioactive molecules, such as pigments, fatty acids, peptides and sterols. Some of these compounds are unique and specifically found in the marine environment and they could be increasingly used as natural bioactive products for targeted applications. Fucoxanthin is one of the major carotenoid found in microalgae well known for its neuroprotective effect but to our knowledge no human studies were realized.

Thus the objective is to evaluate, in healthy older adults, the effect of a 24-week period of daily supplementation of high and low BrainPhyt, doses on cognitive function parameters (Spatial Working Memory scores, Attention and vigilance, episodic memory, executive function), stress, mood, sleep quality and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent and to consume the investigational product daily for the duration of the study.
2. Healthy males and females aged ≥ 55 and ≤ 75 years old.
3. Is free-living (living in a private home, alone or with family, and able to maintain their health and hygiene without assistance).
4. Have age-related mild cognitive decline, defined as:

   1. Absence of dementia as determined by a score of ≥24 on the Mini Mental State Examination (MMSE).
   2. A score on the MAC-Q of ≥25.
5. Have a self-reported memory complaint.
6. Have an AD8 Dementia Screening Score of <2 (normal cognition).
7. Have a Hospital Anxiety and Depression Scale (HADS) score of ≤7 for both anxiety and depression.
8. Is in general good health, as determined by the investigator
9. Ability to comply with study protocol and complete computerised cognitive testing.
10. Willing to maintain their habitual diet and exercise routines.
11. Willing to maintain consistent sleep duration the evening before study visits.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or wish to become pregnant during the study.
2. Female participants currently of childbearing potential, but not using an effective method of contraception, as outlined below:

   1. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where participant discontinues the study prematurely. (Participants utilising this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit).
   2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that participant.
   3. sexual partner(s) is/are exclusively female.
   4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g. male condom, female diaphragm) or contraceptive pill. The participant must be using this method for at least 1 week following the end of the study.
   5. Use of any non-hormonal intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1 % per year. The participant must have the device inserted at least 2 weeks prior to the first Screening Visit, throughout the study, and 2 weeks following the end of the study.
3. Individuals with dementia or mild cognitive impairment defined as greater than or equal to one standard deviation below the mean for age-matched norms on a standardised memory test
4. Individuals taking the following supplements who are unwilling to undergo a 4-week washout period: Ginkgo biloba, Ginseng, Choline, Taurine, Huperizine A, Acetyl-L-Carnitine, DMAE (Dimethylaminoethanol), Lecithin, Phosphatidylcholine, Phosphatidylderine, DHEA (Dehydroepiandrosterene), Alpha lipoic acid, Bacopa (Brahmi), CDP-choline (Citicoline), Alpha-GPC, Green tea extract, L-Tyrosine, or L-Theanine
5. Chronic use of oral or injectable corticosteroids
6. Untreated psychotic or major depressive disorder
7. Uncontrolled hypertension/diabetes
8. A significant history of cardiovascular complaints (e.g., angina)
9. A significant neurological disease
10. Planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study.
11. History within previous 12 months of alcohol or substance abuse.
12. History of heavy smoking (>1 pack/day) within past 3 months.
13. History of heavy caffeinated beverage consumption (>400 mg caffeine/day) within past 2 weeks.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Spatial working memory | From week 0 to week 24
  Change in spatial working memory scores - COMPASS cognitive assessment system

SECONDARY OUTCOMES:
Spatial working memory | From week 0 to week 12
  Change in spatial working memory scores - COMPASS cognitive assessment system
Attention and vigilance | From week 0 to week 24
  Change in spatial working memory scores - COMPASS cognitive assessment system
Attention and vigilance | From week 0 to week 12
  Change in spatial working memory scores - COMPASS cognitive assessment system (Choice reaction time and digit vigilance tasks)
Executive function | From week 0 to week 24
  Change in Executive function scores - COMPASS cognitive assessment system (Stroop task)
Executive function | From week 0 to week 12
  Change in Executive function scores - COMPASS cognitive assessment system (Stroop task)
Episodic memory | From week 0 to week 12
  Change in Episodic memory scores - COMPASS cognitive assessment system (Picture and word recognition tasks)
Episodic memory | From week 0 to week 24
  Change in Episodic memory scores - COMPASS cognitive assessment system (Picture and word recognition tasks)
Sleep quality | From week 0 to week 24
  Change in Leeds sleep evaluation questionnaire score
Sleep quality | From week 0 to week 12
  Change in Leeds sleep evaluation questionnaire score
Mood state | From week 0 to week 24
  Change in Bond-Lader Mood Rating scale score
Mood state | From week 0 to week 12
  Change in Bond-Lader Mood Rating scale score
Stress state | From week 0 to week 24
  Change in Cohen's Perceived stress scale score
Stress state | From week 0 to week 12
  Change in Cohen's Perceived stress scale score
Blood TNFa level (pg/ml) | From week 0 to week 12 and week 24
  Change in blood TNFa compared to baseline
Blood IFN level (pg/ml) | From week 0 to week 12 and week 24
  Change in blood IFN compared to baseline
Blood CRP level (pg/ml) | From week 0 to week 12 and week 24
  Change in blood CRP compared to baseline
Blood IL6 level (pg/ml) | From week 0 to week 12 and week 24
  Change in blood IL6 compared to baseline
Blood Insulin level (mUI/l) | From week 0 to week 12 and week 24
  Change in blood Insulin compared to baseline
Blood HbA1C level (%) | From week 0 to week 12 and week 24
  Change in blood HbA1C compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Professor, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Clinical Food trial, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goodbody E, Maury J, Doolan A, DunnGalvin G, Kakilla C, Pradelles R, Dinan TG. Promising benefits of six-month Phaeodactylum tricornutum microalgae supplementation on cognitive function and inflammation in healthy older adults with age-associated memory impairment. Front Aging. 2025 Apr 30;6:1540115. doi: 10.3389/fragi.2025.1540115. eCollection 2025. PMID 40370669